CLINICAL TRIAL: NCT00115960
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of HIV-1 Gag DNA Vaccine Alone or With IL-15 DNA, Boosted With HIV-1 Gag DNA + IL-15 DNA or HIV-1 Gag DNA + IL-12 DNA, in Healthy, HIV-1 Uninfected Adult Participants
Brief Title: Safety of and Immune Response to an HIV Preventive Vaccine (HIV-1 Gag DNA Alone or With IL-15 DNA) Given With or Without 2 Different Booster Vaccinations in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HVTN 063; 10058 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: IL-12; IL-15; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (6):
- 1 (Experimental): Group 1 will receive 3 vaccinations of the HIV-1 gag DNA vaccine, or placebo. Vaccinations will be given at Months 0, 1, and 3.
  Interventions: Biological: HIV-1 gag DNA
- 2 (Experimental): Group 2 will receive 3 vaccinations of either the HIV-1 gag DNA vaccine with a low dose of IL-15 adjuvant, or a placebo. Vaccinations will be given at Months 0, 1, and 3.
  Interventions: Biological: HIV-1 gag DNA; Biological: IL-15 DNA adjuvant
- 3 (Experimental): Group 3 will receive 3 vaccinations of either the HIV-1 gag vaccine with a medium dose of IL-15 adjuvant, or a placebo. Vaccinations will be given at Months 0, 1, and 3.
  Interventions: Biological: HIV-1 gag DNA; Biological: IL-15 DNA adjuvant
- 4 (Experimental): Group 4 will receive 3 vaccinations of either the HIV-1 gag vaccine with a high dose of IL-15 adjuvant, or a placebo. Vaccinations will be given at Months 0, 1, and 3.
  Interventions: Biological: HIV-1 gag DNA; Biological: IL-15 DNA adjuvant
- 5 (Experimental): In Part B, Group 5 will receive 5 vaccinations of either the HIV-1 gag vaccine plus IL-15 DNA, or placebo. Vaccinations will occur at Months 0, 1, 3, 6, and 9.
  Interventions: Biological: HIV-1 gag DNA; Biological: IL-15 DNA adjuvant
- 7 (Experimental): In Part B, Group 7 will receive 3 vaccinations of the HIV-1 gag vaccine with a high dose of IL-15 adjuvant (maximum tolerated dose from Part A) followed by 2 vaccinations of the gag DNA vaccine with IL-12 DNA adjuvant. Some participants will receive placebo instead of this vaccine regimen. For Group 7, the HIV-1 gag vaccine with IL-15 adjuvant vaccinations will be given at Months 0, 1, and 3, and booster vaccinations will be given at Months 6 and 9.
  Interventions: Biological: HIV-1 gag DNA; Biological: IL-15 DNA adjuvant; Biological: IL-12 DNA adjuvant

INTERVENTIONS:
Biological: HIV-1 gag DNA — DNA vaccine containing the HIV gene gag
Biological: IL-15 DNA adjuvant — Cytokine injection
  Arms: 2; 3; 4; 5; 7
Biological: IL-12 DNA adjuvant — Cytokine injection
  Arms: 7

SUMMARY:
The purpose of this study is to determine the safety of and immune response to an experimental HIV vaccine, HIV-1 gag DNA, with and without an IL-15 DNA adjuvant (at escalating doses of 100, 500, and 1500 mcg). This study will also test the safety of and immune response to the HIV-1 gag DNA vaccine plus IL-15 DNA adjuvant given with or without 2 other adjuvant-containing booster vaccines.

DETAILED DESCRIPTION:
The HIV epidemic is a major global health challenge, causing tremendous human suffering and economic loss throughout the world. The need for a safe, effective, and affordable HIV preventive vaccine is critical. This 2-part study will determine the safety and immunogenicity of the experimental HIV vaccine HIV-1 gag DNA with or without IL-15 adjuvant, boosted with either the HIV-1 gag DNA and IL-15 adjuvant vaccine or the HIV-1 gag DNA and IL-12 adjuvant vaccine.

There are two parts to this study. Part A will last 12 months. In Part A, 48 participants will be randomly assigned to 1 of 4 groups in sequential order (dose escalation). All participants will receive 3 vaccinations. Group 1 will receive 3 vaccinations of the HIV-1 gag DNA vaccine or placebo. Group 2 will receive 3 vaccinations of either the HIV-1 gag DNA vaccine with a low dose of IL-15 adjuvant or a placebo. Group 3 will receive 3 vaccinations of either the HIV-1 gag vaccine with a medium dose of IL-15 adjuvant or a placebo. Group 4 will receive 3 vaccinations of either the HIV-1 gag vaccine with a high dose of IL-15 adjuvant or a placebo. Vaccinations will be given at Months 0, 1, and 3. There will be 11 study visits in Part A. A physical exam, pregnancy prevention counseling, medication history, and adverse event reporting will occur at most visits. Urine and blood collection will occur at some visits. Participants will also be asked to complete questionnaires at certain visits.

Part B will last 15 months. In Part B, 72 participants will be randomly assigned to 1 of 2 groups. All Part B participants will receive 5 vaccinations. Group 5 will receive 5 vaccinations of either the HIV-1 gag vaccine plus IL-15 DNA or placebo; the vaccinations will occur at Months 0, 1, 3, 6, and 9. Group 7 will receive 3 vaccinations of the HIV-1 gag vaccine with a high dose of IL-15 adjuvant (maximum tolerated dose from Part A) followed by 2 vaccinations of the gag DNA vaccine with IL-12 DNA adjuvant. Some participants will receive placebo instead of this vaccine regimen. For Group 7, the HIV-1 gag vaccine with IL-15 adjuvant vaccinations will be given at Months 0, 1, and 3, and booster vaccinations will be given at Months 6 and 9. There will be 13 study visits in Part B. A physical exam, pregnancy prevention counseling, medication history, and adverse event reporting will occur at most visits. Urine and blood collection will occur at some visits. Participants will also be asked to complete questionnaires at certain visits.

ELIGIBILITY:
Note: Group 6 has been removed from Part B of the protocol as of the 04/11/06 amendment. Because a regimen similar to Group 6's regimen is being tested in HVTN 060, the vaccine manufacturer decided that Group 6's regimen was not a priority for testing.

Inclusion Criteria:

* HIV uninfected
* Access to a participating HIV Vaccine Trials Unit (HVTU)
* Willing to receive HIV test results
* Willing and able to comply with all study requirements
* In good general health
* Willing to use acceptable methods of contraception for at least 21 days prior to study entry and until the last study visit. More information about this criterion can be found in the protocol.
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus (anti-HCV) antibody negative or negative HCV PCR if anti-HCV antibody is positive

Exclusion Criteria:

* HIV vaccines in prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to first vaccination
* Blood products within 120 days prior to first vaccination
* Immunoglobulin within 60 days prior to first vaccination
* Live attenuated vaccines within 30 days prior to first vaccination
* Investigational research agents within 30 days prior to first vaccination
* Medically indicated subunit or killed vaccines within 14 days prior to first study vaccine administration, or allergy treatment with antigen injections within 30 days prior to first vaccination
* Current tuberculosis (TB) prophylaxis or therapy
* Clinically significant medical condition, physical exam findings, abnormal laboratory results, or past medical history with clinically significant implications for current health
* Any medical, psychiatric, or social condition that, in the opinion of the investigator, may interfere with the study
* Any occupational or other responsibility that, in the opinion of the investigator, may interfere with the study
* Diagnosis of allergy to amide-type local anesthetics
* Serious adverse reaction to vaccines, including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, or abdominal pain. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Unstable asthma
* Diabetes mellitus Type 1 or Type 2. Participants with histories of isolated gestational diabetes are not excluded.
* Thyroid disease requiring treatment in the past 12 months
* Serious angioedema within the last 3 years
* Uncontrolled hypertension
* Body mass index (BMI) of 40 or greater OR BMI of 35 or greater, when certain other criteria are met. More information about these criteria can be found in the protocol.
* Bleeding disorder
* Cancer. Participants with surgically removed cancer that, in the opinion of the investigator, is unlikely to recur are not excluded.
* Seizure disorder requiring medication within the past 3 years
* Absence of the spleen
* Psychiatric condition, including psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years
* Pregnant or breastfeeding, or plan to become pregnant during the study

Exclusion Criteria for Part B Participants:

* Diagnosis of allergy to egg products
* Diagnosis of allergy to yeast-derived products

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Local and systemic reactogenicity signs and symptoms, as assessed after each injection | 12 months postinjection for Part A, and 15 months after the first injection in Part B
Laboratory measures of safety, as assessed after each injection | 12 months postinjection for Part A, and 15 months after the first injection in Part B
Adverse and serious adverse experiences, as assessed after each injection | 12 months postinjection for Part A, and 15 months after the first injection in Part B

SECONDARY OUTCOMES:
HIV-specific cellular responses by IFN-gamma ELISpot | 12 months postinjection for Part A, and 15 months after the first injection in Part B
HIV binding antibody by ELISA | 12 months postinjection for Part A, and 15 months after the first injection in Part B
Social impact variables | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, MD, Study Chair — Harvard University; Xia Jin, MD, PhD, Study Chair — University of Rochester
Locations (7):
- United States (6):
  - Brigham and Women's Hosp. CRS, Boston, Massachusetts
  - NY Blood Ctr./Union Square CRS, New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - NY Blood Ctr./Bronx CRS, The Bronx, New York
  - Miriam Hospital's HVTU, Providence, Rhode Island
- Sao Paulo HVTU - CRT DST/AIDS CRS, São Paulo, Brazil

REFERENCES:
- [Background] Boyer JD, Chattergoon M, Muthumani K, Kudchodkar S, Kim J, Bagarazzi M, Pavlakis G, Sekaly R, Weiner DB. Next generation DNA vaccines for HIV-1. J Liposome Res. 2002 Feb-May;12(1-2):137-42. doi: 10.1081/lpr-120004786. PMID 12604047
- [Background] Stratov I, DeRose R, Purcell DF, Kent SJ. Vaccines and vaccine strategies against HIV. Curr Drug Targets. 2004 Jan;5(1):71-88. doi: 10.2174/1389450043490686. PMID 14738219
- [Background] Xin KQ, Hamajima K, Sasaki S, Tsuji T, Watabe S, Okada E, Okuda K. IL-15 expression plasmid enhances cell-mediated immunity induced by an HIV-1 DNA vaccine. Vaccine. 1999 Feb 26;17(7-8):858-66. doi: 10.1016/s0264-410x(98)00271-0. PMID 10067692
- [Derived] Jin X, Morgan C, Yu X, DeRosa S, Tomaras GD, Montefiori DC, Kublin J, Corey L, Keefer MC; NIAID HIV Vaccine Trials Network. Multiple factors affect immunogenicity of DNA plasmid HIV vaccines in human clinical trials. Vaccine. 2015 May 11;33(20):2347-53. doi: 10.1016/j.vaccine.2015.03.036. Epub 2015 Mar 25. PMID 25820067
- [Derived] Kalams SA, Parker S, Jin X, Elizaga M, Metch B, Wang M, Hural J, Lubeck M, Eldridge J, Cardinali M, Blattner WA, Sobieszczyk M, Suriyanon V, Kalichman A, Weiner DB, Baden LR; NIAID HIV Vaccine Trials Network. Safety and immunogenicity of an HIV-1 gag DNA vaccine with or without IL-12 and/or IL-15 plasmid cytokine adjuvant in healthy, HIV-1 uninfected adults. PLoS One. 2012;7(1):e29231. doi: 10.1371/journal.pone.0029231. Epub 2012 Jan 5. PMID 22242162